CLINICAL TRIAL: NCT02227381
Title: Using New Genetic Technology to Diagnose Neurodevelopmental Disorders
Brief Title: Action Medical Research
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 10/H1003/98; SP4555 (Other Grant/Funding Number: Action Medical Research)
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Learning Disabilities
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from whole blood, saliva or skin biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Microarray / NGS test

SUMMARY:
Learning disability affects 3% of the population. Severe types of learning disability are more likely to have an underlying genetic cause but diagnosis is difficult because many different genetic abnormalities may be involved. Obtaining a diagnosis is important so that patients can be managed appropriately and their families can be given accurate information.

We aim to use new types of genetic testing which will make it possible to screen for several different genetic abnormalities which cause learning disability at the same time, so improving the accuracy and speed of diagnosis in the group of patients with severe learning disability. We will focus particularly on patients where seizures and behavioural problems are also present.This will enable more patients to be diagnosed accurately, reduce the number of hospital appointments needed and ultimately be more cost- effective.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with severe learning disability associated with either seizures, movement or behaviour problems who had previously undergone routine investigation but where no cause had been identified for their problems

Exclusion Criteria:

* Individuals with SLD where the cause is already known
* Individuals where informed consent cannot be obtained for participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will approach a cohort of patients with severe LD/seizures/behaviour problems who have presented to us in our genetic clinic for diagnosis over the past few years, but where the cause of their problems remains unknown. This will be our study population. In virtually all cases we will have performed routine diagnostic testing and will have stored DNA.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Genetic abnormality identified by microarray or Next Generation Sequencing | up to 6 months following consent
  Abnormalities identified upon results of testing, the normal timeframe for this is up to 6 months after collecting blood sample.

SECONDARY OUTCOMES:
Cost effectiveness vs normal care | By the end of the study (December 2014)
  This analysis will be performed for all participants following close of recruitment & follow up, and will be completed by the time the study ends.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Clayton Smith, MB ChB FRCP MD, Principal Investigator — CMFT
Locations (1):
- Central Manchester University Hospitals NHS Foundation Trust, Manchester, United Kingdom